CLINICAL TRIAL: NCT02119871
Title: Comparative Effectiveness of Unilateral Versus Bilateral Pulmonary Collapse in De-airing During Open Left Heart Surgery.
Brief Title: Comparative Effectiveness of Unilateral vs. Bilateral Pulmonary Collapse in Cardiac De-airing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Bansi Lal Koul, Lund University, Lund University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BKML-004
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Results first posted 2018-01-29 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2017-06

CONDITIONS: Brain Ischemia; Reduction of Cerebral Air Emboli
Keywords: Cerebral air emboli, heart surgery
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bilateral Open Pleurae (Experimental): Bilateral open pleurae and usage of right pulmonary vein drainage
  Interventions: Procedure: Bilateral Open Pleurae
- Right pleura open (Active Comparator): Opening of right pleura and usage of left ventricular apical drainage.
  Interventions: Procedure: Right Pleura Open

INTERVENTIONS:
Procedure: Bilateral Open Pleurae — Both pleurae are opened Right pulmonary vein drainage
  Arms: Bilateral Open Pleurae
Procedure: Right Pleura Open — Right pleura open Left ventricular apical drainage
  Arms: Right pleura open

SUMMARY:
To compare the effectiveness of unilateral pulmonary collapse (right lung) to bilateral pulmonary collapse for cardiac de-airing in open left-sided heart surgery.

DETAILED DESCRIPTION:
Effective removal of air from the heart before termination of cardiopulmonary bypass (CPB) is vital in open left heart surgery. Bilateral collapse of the lungs during cardiopulmonary bypass decreases the duration of the de-airing procedure, decreases residual air emboli monitored on Trans-esophageal Echocardiography (TEE) and decreases gaseous cerebral microemboli (MES) monitored by Trans-cranial Echo-Doppler (TCD) when compared to expanded lungs during (CPB). Induced pulmonary collapse by opening of the pleura and disconnection of the patient from the ventilator during CPB decreases the amount of air that can enter the pulmonary veins. Not all surgeons wish to induce lung collapse from fraught that it might lead to pulmonary ischemia or infection. It is unknown whether collapse of only the right lung is as effective as collapse of both lungs.

ELIGIBILITY:
Inclusion Criteria:

* Aortic valve pathology requiring surgery.

Exclusion Criteria:

* Prior thoracic surgery,
* Severe chronic obstructive pulmonary disease and/or
* Emphysema.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bansi Koul, MD, PhD, Principal Investigator — Lund University
Locations (1):
- Department of Cardiothoracic Department, Skane University Hospital, Lund, Lund, Skåne, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who were scheduled for elective open left heart surgery at Skåne University Hospital were eligible for inclusion.
Period: Overall Study
Arm/Group | Bilateral Open Pleurae | Right Pleura Open
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Groups were statistically compared to a historical control group of 10 patients with bilateral open pleurae and left ventricular apical vent.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bilateral Open Pleurae | Right Pleura Open | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69 [65 to 74] | 71 [64 to 79] | 70 [65 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 7 | 6 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 10 | 10 | 20
Body surface area [Median (Inter-Quartile Range); unit: m^2] | 1.97 [1.71 to 2.13] | 1.93 [1.79 to 2.11] | 1.97 [1.79 to 2.11]

OUTCOME MEASURES:

1. Primary Outcome: Quantitative Assessment of Air Embolism to the Brain After Completion of Open Left Heart Surgery
Description: Cerebral air emboli will be assessed quantitatively by On-line counting of gaseous microembolic signals (MES) by Trans-cranial Echo-Doppler (TCD) monitoring of the right and left middle cerebral artery. The sum of the gaseous microembolic signals registered from the right and the left middle cerebral artery will be reported.
Time Frame: Time from the release of the aortic crossclamp to cardiac ejection, an average of 5-10 minutes
Population: Groups were statistically compared to a historical control group of 10 patients with bilateral open pleurae and left ventricular apical vent (LVAV) in order to evaluate:1. the impact on de-airing of unilateral open pleura compared to bilateral open pleurae, and 2. the impact on de-airing of a right superior pulmonary vein vent compared to LVAV.
Measure: Median (Inter-Quartile Range); unit: gaseous cerebral microemboli
Arm/Group | Bilateral Open Pleurae | Right Pleura Open
Number analyzed (Participants) | 10 | 10
gaseous cerebral microemboli | 46 [21 to 107] | 32 [16 to 68]
Statistical Analysis 1: Comparison: Bilateral Open Pleurae vs Right Pleura Open; Test type: Superiority; p = 1.00, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 14

2. Primary Outcome: Quantitative Assessment of Air Embolism to the Brain After Completion of Open Left Heart Surgery
Description: as for outcome 1
Time Frame: Time from cardiac ejection to finished de-airing, an average on 5-10 minutes
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: gaseous cerebral microemboli
Arm/Group | Bilateral Open Pleurae | Right Pleura Open
Number analyzed (Participants) | 10 | 10
gaseous cerebral microemboli | 31 [10 to 166] | 41 [27 to 55]
Statistical Analysis 1: Comparison: Bilateral Open Pleurae vs Right Pleura Open; Test type: Superiority; p = 0.656, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 10

3. Primary Outcome: Quantitative Assessment of Air Embolism to the Brain After Completion of Open Left Heart Surgery
Description: as for outcome 1
Time Frame: Period of ten minutes after finished de-airing
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: gaseous cerebral microemboli
Arm/Group | Bilateral Open Pleurae | Right Pleura Open
Number analyzed (Participants) | 10 | 10
gaseous cerebral microemboli | 30 [9 to 75] | 34 [14 to 43]
Statistical Analysis 1: Comparison: Bilateral Open Pleurae vs Right Pleura Open; Test type: Superiority; p = 1, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 4

4. Primary Outcome: Number of Participants With <=Grade I Air Emboli as Assessed by Trans-esophageal Echocardiography (TEE) After Finished De-airing.
Description: The severity of residual air emboli in three anatomic areas; left atrium, left ventricle and the aortic root, is assessed by Trans-esophageal Echocardiography (TEE) and classified in grade 0-3 as follows: Grade 0: no residual air emboli, Grade I: air emboli observed in one of three anatomic areas, Grade II: air emboli observed simultaneously in two of three anatomic areas, Grade III: air emboli observed simultaneously in all three anatomic areas.
Time Frame: 0-3 minutes after finished de-airing
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Bilateral Open Pleurae | Right Pleura Open
Number analyzed (Participants) | 10 | 10
Participants | 8 | 9

5. Primary Outcome: Number of Participants With <=Grade I Air Emboli as Assessed by Trans-esophageal Echocardiography (TEE) After Finished De-airing.
Description: as for outcome 4
Time Frame: 3-6 minutes after finished de-airing
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Bilateral Open Pleurae | Right Pleura Open
Number analyzed (Participants) | 10 | 10
Participants | 9 | 10

6. Primary Outcome: Number of Participants With <=Grade I Air Emboli as Assessed by Trans-esophageal Echocardiography (TEE) After Finished De-airing.
Description: as for outcome 4
Time Frame: 7-10 minutes after finished de-airing
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Bilateral Open Pleurae | Right Pleura Open
Number analyzed (Participants) | 10 | 10
Participants | 9 | 10

7. Secondary Outcome: Duration of the De-airing Procedure
Description: Duration of the de-airing procedure counted in minutes.
Time Frame: Duration in minutes fråm removal of the aortic cross clamp to finished de-airing, an average of 10-15 minutes.
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Bilateral Open Pleurae | Right Pleura Open
Number analyzed (Participants) | 10 | 10
minutes | 8 [6 to 12] | 10 [7 to 11]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the inpatient care period after surgery, approximately 1 week.
Arm/Group | Bilateral Open Pleurae | Right Pleura Open
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bilateral Open Pleurae (N=10) | Right Pleura Open (N=10)
Neurological deficit (Nervous system disorders) | 1 (1) | 1 (1) — Any type of postoperative transient or permanent neurological dysfunction detected at routine bedside investigation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes